CLINICAL TRIAL: NCT00317226
Title: Open Label Extension Study Evaluating the Long Term Safety, Tolerability and Efficacy of an Iron Maintenance Dosing Strategy Utilizing Intravenous VIT45 in the Treatment of Anemia in Non-Dialysis Dependent Chronic Kidney Disease
Brief Title: Long Term Safety Study of (VIT45) Extension Study: Treatment of Anemia in Non-Dialysis Dependent Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT05005
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
Keywords: Anemia; CKD; Chronic Kidney Disease; Iron; Maintenance Dose
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferric Carboxymaltose (FCM) (Experimental): maximum dose of 1,000 mg over 15 minutes IV administered within 7 days of the qualifying visit
  Interventions: Drug: Ferric Carboxymaltose (FCM)

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — maximum dose of 1,000 mg over 15 minutes IV administered within 7 days of the qualifying visit

SUMMARY:
The primary objective of this study is to evaluate the long term safety and tolerability of an iron maintenance dosing strategy utilizing VIT45 in the treatment of anemia of non-dialysis dependent chronic kidney disease (NDD-CKD). This study is a long term extension to protocol 1VIT04004 (NCT00317239).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the long term safety and tolerability of an iron maintenance dosing strategy utilizing VIT45 in the treatment of anemia of non-dialysis dependent chronic kidney disease (NDD-CKD). This study is a long term extension to protocol 1VIT04004.

In this study patients that complete protocol 1VIT 04004 or are discontinued will be offered to participate in this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed or discontinued Protocol 1VIT04004

Exclusion Criteria:

* Known hypersensitivity reaction to VIT-45
* Anemia not related to CKD
* Chronic, serious infection
* Recent IV iron other than study drug in past 12 weeks
* Recent blood loss within the last 12 weeks
* Need for surgery or dialysis
* Female subjects who are pregnant or lactating

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2005-06; Primary Completion 2007-03 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals Inc., Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Pre-assignment Details: no treatment with FCM in the trial excluded 18 subjects from the Safety population
Groups:
- Ferric Carboxymaltose (FCM): maximum dose of 1,000 mg over 15 minutes IV administered within 7 days of the qualifying visit based on TSAT and Ferritin levels
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM)
Started | 127
Completed | 104
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | Ferric Carboxymaltose (FCM)
Number analyzed (Participants) | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 61
  >=65 years | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 127

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events
Time Frame: 44 week study duration
Measure: Number; unit: each event
Arm/Group | Ferric Carboxymaltose (FCM)
Number analyzed (Participants) | 127
each event | 84

ADVERSE EVENTS:
Time Frame: 1 year and 8 months
Arm/Group | Ferric Carboxymaltose (FCM)
Serious Adverse Events (participants affected / at risk) | 23/127
Other Adverse Events (participants affected / at risk) | 23/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=127)
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 2
Localized infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Localized osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Anoxic encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Azotemia (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Carboxymaltose (FCM) (N=127)
Odema peripheral (General disorders) | 9
Urinary tract infection (Infections and infestations) | 7
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less